CLINICAL TRIAL: NCT01407510
Title: A Multicenter, Open-label Study to Evaluate the Adrenal Suppression Potential of Mapracorat 0.1% Ointment in Japanese Adults With Atopic Dermatitis
Brief Title: HPA Axis Study in Japanese Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15519; 1403460 (Other: Company Internal)
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Mapracorat

INTERVENTIONS:
Drug: Mapracorat — Application of the investigational product on the affected skin areas

SUMMARY:
A multicenter, open-label study to evaluate the adrenal suppression potential of Mapracorat 0.1% ointment in Japanese adults with atopic dermatitis.

DETAILED DESCRIPTION:
Assessment of the adrenal suppression potential, safety, efficacy and pharmacokinetics of Mapracorat 0.1% ointment in Japanese adults with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female subject aged >= 20 years
* Diagnosis of atopic dermatitis according to the Hanifin and Rajka criteria
* Investigator's Global Assessment (IGA) score of 3 (moderate) to 4 (severe) at baseline
* Normal ACTH response before start of treatment

Exclusion Criteria:

* Pregnancy or lactation
* Clinically relevant disease, which could interfere with the study conduct or the evaluation and interpretation of the study results
* Concomitant medical or dermatological disorder(s), which could interfere with the investigator's ability to evaluate the subject's response to the investigational product
* Clinically manifest immunosuppressive disorder or known history of malignant disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05-09 (Actual); Primary Completion 2011-09-16 (Actual); Study Completion 2012-04-15 (Actual)

PRIMARY OUTCOMES:
number of subjects with adrenal suppression

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Kawaguchi Kogyo General Hospital, Saitama
  - Clinical Research Hospital Tokyo, Tokyo
  - Tokyo Women's Medical University, Tokyo